CLINICAL TRIAL: NCT06132620
Title: Clinical Efficacy of Qingxin Zishen Decoction in Treating Menopausal Syndrome and Neuroendocrine Mechanism of Regulating KNDy Neurons
Acronym: QXZSKNDy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yun Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Chen, Deputy Chief Physician, Jiangsu Province Hospital of Traditional Chinese Medicine
Organization: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QXZS-1
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Menopause
MeSH Terms: interventions — femoston

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental)
  Interventions: Drug: Qingxin Zishen Decoction
- the control group (Active Comparator)
  Interventions: Drug: Femoston

INTERVENTIONS:
Drug: Femoston — Fenmorphone (this product is a compound preparation, estradiol tablets contain estradiol 2mg; Estradiol dydrogesterone tablets contain estradiol 2 mg and dydrogesterone 10 mg).
  Usage: 1 time/day: 1 tablet orally every day, every 28 days as a course of treatment.
  Arms: the control group
Drug: Qingxin Zishen Decoction — Qingxin Zi Kidney Decoction is a traditional Chinese medicine decoction, after regular decoction, 1 dose/day, divided into 2 doses.
  Arms: the experimental group

SUMMARY:
The goal of this clinical trial is to determine the effects of estrogen (Fenmotong) and Qingxin Zishen Decoction on the levels of kisspeptin, NKB, and dynorphin expressed in human KNDy neurons Between patients with menopausal syndrome. The aims of the study are as follows:

* Find a new neuroendocrine mechanism of Qingxin Zishen Decoction in the treatment of menopausal syndrome.
* Evaluate the changes of new neuroendocrine indicators in the clinical treatment of menopausal syndrome.
* Develop non-hormonal drugs with definite efficacy in the treatment of menopausal syndrome.

Participants will randomly divided into the experimental group and the control group, the experimental group will be oral fenmotong, and the control group will be oral Qingxin Zi Kidney Decoction, and the efficacy, sex hormone levels and neuroendocrine index changes of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 41~55;
* KIM score≥ 15 points;
* The number of hot flashes and sweating≥ 3 times/day;
* Menopause time≥ 6 months;
* FSH>30mIU/ml,E2<30ng/L;
* Informed consent, voluntary testing.

Exclusion Criteria:

* Unexplained vaginal bleeding;
* Sex hormone-related malignant tumors cannot be excluded;
* premature ovarian failure, or endometriosis, or hysterectomy, or bilateral adnexectomy;
* Combined with primary liver and kidney dysfunction, cardiovascular and cerebrovascular diseases, blood system diseases and other serious diseases that affect their survival;
* Exposure to sex hormone-related drugs within 3 months;
* Patients with mental abnormalities, or those with a history of alcohol or drug abuse;
* Those who have allergic reactions to the study drug;
* Those who are participating in other drug clinical researchers.

Ages: 41 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Modified Kupperman Menopausal Index | Baseline, at the 4th, 8th and 12th weeks of treatment
  The Modified Kupperman Menopausal Index is a scoring method to evaluate women's menopausal related symptoms, using the Kupperman index (KMI) score, including 13 menopausal related symptoms such as vasomotor symptoms, paresthesias, and insomnia ...Each symptom is divided into 0 to 3 points according to severity, and multiplied by different coefficients to obtain the menopausal symptom index, when the index > 35 indicates severe symptoms, 21-35 indicates moderate symptoms, and 15-20 indicates mild symptoms.
Hot flashes and sweats on a five-level scale | Baseline, at the 4th, 8th and 12th weeks of treatment
  The symptoms of hot flashes and sweating were recorded as none, mild, moderate, severe, and very severe, and were recorded as 0, 1, 2, 3, and 4 points. Higher scores indicate more severe symptoms.
sex hormone | Baseline and 12th weeks of treatment
  Patients who met the inclusion criteria were collected 5 ml of cubital venous blood on an empty stomach before and after treatment, and serum estradiol (E2) and follicle-stimulating hormone (FSH) levels were detected by chemiluminescence method.
Neuroendocrine indicators | Baseline and 12th weeks of treatment
  The patients who met the inclusion criteria were fasted before and after treatment, and the levels of hypothalamic neuronal active peptide (kisspeptin), neurokinin B (NKB) and dynorphin (Dyn) were detected by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Yuxin Zhou, Nanjing, 南京, China

IPD SHARING:
Plan to Share IPD: No